CLINICAL TRIAL: NCT06560879
Title: Effectiveness of Probiotics for the Prevention of Gastrointestinal Toxicity and Changes in Gut Microbiota in Children with Acute Lymphoblastic Leukemia
Brief Title: Effectiveness of Probiotics for the Prevention of Gastrointestinal Toxicity in Children with Leukemia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Pediatrics, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021/030
Record Dates: First submitted 2024-08-06; First posted 2024-08-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-11

CONDITIONS: Probiotics; Gastrointestinal Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Gastrointestinal Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: An experimental, longitudinal, prospective, prolective, analytical, concurrent, randomized, triple-blind: randomized controlled clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Interventions packaged in identical, odorless, tasteless, opaque capsules; stored in identical white plastic bottles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Lactobacillus casei (Experimental): Oral administration of 1 capsule with Lactobacillus casei (2.5 billion CFU + microcrystalline cellulose) before breakfast and another capsule before lunch, for a total dose of 5 billion CFU/day.
  Interventions: Biological: Lactobacillus casei
- Lactobacillus rhamnosus (Experimental): Oral administration of 1 capsule with Lactobacillus rhamnosus (2.5 billion CFU + microcrystalline cellulose) before breakfast and another capsule before lunch, for a total dose of 5 billion CFU/day.
  Interventions: Biological: Lactobacillus rhamnosus
- Bifidobacterium bifidum (Experimental): Oral administration of 1 capsule with Bifidobacterium bifidum (1 billion CFU + microcrystalline cellulose) before breakfast and another capsule before lunch, for a total dose of 2 billion CFU/day.
  Interventions: Biological: Bifidobacterium bifidum
- Placebo (Placebo Comparator): Oral administration of 1 capsule of 300 mg of microcrystalline cellulose before breakfast and another before lunch (600 mg/day).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Biological: Lactobacillus casei — Lacticaseibacillus casei is a species of Gram-positive anaerobic bacteria found in the intestine and mouth of humans. This lactic acid-producing bacterium is used in the dairy industry in the production of probiotic foods.
  Arms: Lactobacillus casei
Biological: Lactobacillus rhamnosus — A live form of a bacterium that makes lactic acid (a substance derived from milk sugars and also made by the body). Lactobacillus rhamnosus GG is given to help with digestion and normal bowel function. In addition, it may help maintain a healthy gastrointestinal tract. It is being studied for the prevention of infections in patients who received donor stem cell transplants and for other conditions.
  Arms: Lactobacillus rhamnosus
Biological: Bifidobacterium bifidum — B. bifidum is an essential bacteria found in the human intestine. When it is low or absent all together in the human intestine, it is an indication of being in an unhealthy state. Intestinal flora can be improved if someone takes oral B. bifidum. Also, oral B. bifidum is used for other things such as therapy for enteric and hepatic disorders, for activating the immune response, and for preventing some cancers
  Arms: Bifidobacterium bifidum
Dietary Supplement: Placebo — Microcrystalline cellulose is a term for refined wood pulp and is used as a texturizer, an anti-caking agent, a fat substitute, an emulsifier, an extender, and a bulking agent in food production.The most common form is used in vitamin supplements or tablets
  Arms: Placebo

SUMMARY:
Background: Acute lymphoblastic leukemia (ALL) is a common malignant neoplasm in children. Although chemotherapy achieves remission in over 70% of cases, it can cause gastrointestinal toxicity in up to 32.5%. Some studies suggest that administering probiotics reduces this risk, but the evidence remains inconsistent.

Objective: To evaluate the effectiveness and safety of administering L. casei, L. rhamnosus or B. bifidum compared to a placebo for the prevention of gastrointestinal toxicity, decreased intestinal permeability, and changes in intestinal microbiota in pediatric patients diagnosed with acute lymphoblastic leukemia receiving chemotherapy.

Methods: A total of 120 participants aged 6 to 17 years, diagnosed with ALL and receiving consolidation phase chemotherapy without gastrointestinal comorbidities, will be included. Participants will be administered daily 2 capsules containing either 1) L. casei, 2) L. rhamnosus, 3) B. bifidum or 4) placebo daily for 8 weeks. The clinical status of the participants will be evaluated weekly by the oncology service to determine the presence of gastrointestinal toxicity and adverse events. Changes in intestinal permeability will be assessed by measuring beta-lactoglobulin in a blood sample using the ELISA technique, while changes in the intestinal microbiota will be analyzed by genomic sequencing at baseline and at the end of follow-up.

Statistical analysis: Descriptive analysis will use measures of central tendency and dispersion. For quantitative variables, the mean and standard deviation or median with minimum and maximum values will be calculated depending on the distribution type. Frequencies and proportions will be calculated for qualitative variables, presented in tabular and graphical form. To compare the quantitative variables between the four interventions, a multi-way ANOVA test will be used.

The risk of gastrointestinal toxicity and adverse events will be analyzed by calculating the relative risk and 95% confidence interval. Differences between the interventions will be analyzed using survival analysis with the Kaplan-Meier and Log-Rank tests. Sequencing data will be analyzed using the Qiime2 program, filtered to generate a phylogenetic tree using the Silva database. Corresponding plots will be generated for each taxonomic level. Alpha (intra-group) and Beta (inter-group) diversity will be presented by ordination plots using principal component analysis with the ANCOM program

DETAILED DESCRIPTION:
Background Acute lymphoblastic leukemia (ALL) is a malignant disease characterized by the uncontrolled proliferation of immature lymphoid cells. It is the most common neoplasm in children, representing up to 53.1% of all oncologic processes in Mexico [1-6]. Fortunately, with the current chemotherapeutic treatments, disease remission is achieved in 98% of cases; however, the chemotherapeutic treatments have side effects that can lead to gastrointestinal toxicity (7.7 to 32.5%), which is associated with up to 50% mortality.

Among the most common gastrointestinal manifestations resulting from this toxicity are mucositis, pancreatitis (2 to 8%), diarrhea (10 to 82%), and colitis associated with decreased Bacillus spp and Bidifobacterium spp, increasing the risk of necrosis and intestinal perforation of the terminal ileum and cecum. Hence, several studies have been conducted to identify agents that can reduce the incidence of gastrointestinal toxicity like as probiotics which are a group of saprophytic microorganisms (bacteria, viruses, fungi and protozoa) that live in equilibrium on the skin and mucous membranes, mainly in the intestine, have garnered attention.

Probiotics are known to have several beneficial functions such as promoting the absorption of carbohydrates, short-chain fatty acids and calcium; facilitating the synthesis of lipids and vitamins; modulate and reduce the concentration of inflammatory mediators in the intestinal mucosa; improve mucosal blood flow, thus reducing the risk of ischemic areas in the intestine; and strengthen the immune system.

Although research has been conducted on the use of probiotics to prevent or reduce the toxic effects of chemotherapy, the results are still inconclusive because the effect of probiotics has been analyzed in multiple combinations, which makes it difficult to distinguish the specific effects per phylum. This complicates the generation of standardized therapeutic schemes to improve the quality of care of these patients. If this project successfully identifies the effectiveness and safety of these probiotics, it will enable to development of new therapeutic strategies aimed at improving the quality of healthcare for these patients, reducing the frequency and severity of gastrointestinal complications secondary to the administration of chemotherapy.

Objective To evaluate the effectiveness and safety of the administration of Lactobacillus casei, Lactobacillus rhamnosus and Bifidobacterium bifidum compared to placebo in reducing the risk of gastrointestinal toxicity, decreasing intestinal permeability, and changing intestinal microbiota without the development of adverse effects in pediatric patients diagnosed with ALL receiving consolidation chemotherapy in the Oncology Service of the Instituto Nacional de Pediatría.

General Description of the Study

1. Participant selection and consent:

   * Participants meeting the study selection criteria will be selected.
   * Informed consent will be obtained from the participant's parents or guardians and, if appropriate, from the patient if older than 8 years of age. They will be informed about the benefits, complications and adverse effects of the interventions (Appendix 1-3).
   * If the parents or guardians prefer treatment outside the research project, the patient will be treated according to the established national protocols used in the Oncology Service of the Instituto Nacional de Pediatría.
   * Consent will also be obtained for the use of personal data as per Appendices 4 and 5. This data includes participant and parent names, birth date, sex, CURP, address, contact number, medical history, general habits, pathological conditions, social conditions, to be used exclusively for this research project.
   * Data will be handled with strict confidentiality, stored in an electronic database for five years by project personnel.
2. Initial Assessments:

   * A pediatric oncologist will perform a medical history, physical examination, anthropometry, fecal and serum sampling.
   * A nutritionist will evaluate the participant´s nutritional status and body composition.

   A) Physical examination:
   * Participant will remove outer clothing and shoes and sit on the examination table.
   * The pediatric oncologist will visually inspect for skin lesions using a lamp and tongue depressor if necessary.
   * Body temperature will be measured with a digital thermometer.
   * Participants will lie supine for palpation, percussion, and/or auscultation to assess cardiac, and abdominal conditions.

   B) Anthropometry
   * Weight will be measured three times using a Seca scale.
   * Height will be measured three times using a stadiometer.
   * Waist circumference will be measured at the midpoint between the lower edge of the last rib and the upper edge of the iliac crest.
   * Hip circumference will be measured 15 cm below the waist.
   * Arm circumference will be measured around the biceps muscle.
   * Thigh circumference will be measured around the upper third of the thigh.

   C) Nutritional Status

   - Height-for-Age (H-A), Weight-for-Age (W-A), Weight-for-Height (W-H), and Body Mass Index (BMI) indices will be classified according to NOM-008-SSA2-1993 standards.

   D) Body composition
   * Participants will remove metallic objects, empty their bladder, and lie supine on a non-conductive bed.
   * Electrode placement will be prepared with a cleansing towel and an electrically conductive towel.
   * Electrodes will be placed on hands and feet, and a multifrequency bioelectric impedance device will measure body composition at six different frequencies.
   * Data will be adjusted to WHO percentile curves.

   E) Fecal samples
   * Participants will collect stool samples at home using provided kits and instructions.
   * Samples will be transported in a cooler to the Instituto Nacional de Pediatría on the same day for analysis and will be stored in the freezer at -70°C until the end of the project.

   F) Serum samples
   * A 3 ml blood sample will be collected by peripheral venipuncture.
   * Serum samples will be processed to determine antibodies against beta-lactoglobulin using the sandwich enzyme immunoassay technique.

   Assessments will be conducted weekly for clinical condition, anthropometry, and body composition at weeks 1, 4, and 8, and fecal and serum samples at weeks 1 and 8.
3. Preparation of interventions:

   * Interventions will be prepared in a Baker Company Class II Type A2 vertical laminar flow hood.
   * The required amounts of lyophilized probiotic powder and microcrystalline cellulose will be mixed for 5 minutes (2:30 clockwise and 2:30 counterclockwise) at a speed of 25 rpm and encapsulated at a dose of: L. casei and L. rhamnosus at 2.5 billion CFU per capsule, B. bifidum at 1 billion CFU per capsule and placebo 300 mg of microcrystalline cellulose.
   * Each intervention will be stored in labeled sterile bags and refrigerated at 2 to 8°C.
   * Capsules will be quality checked for UFC content at Bacteriology Laboratory by dilution and sequencing, and any deviations will result in process adjustments.
4. Participant Allocation:

   * Participants will be randomly assigned to interventions using a computer-generated sequence, adjust in balanced blocks of five. (Appendix 7).
   * An external researcher will place intervention names in opaque envelopes, labeled with random numbers of the sequence.
   * Participants will draw a random number to be assigned to an intervention, communicated to the principal investigator.
5. Intervention Administration:

   * Participants will receive bottles with 14-16 capsules of the assigned intervention, stored in a cooler with refrigerated gel packs.
   * Participants will take one capsule before breakfast and one before lunch for one week, recording adherence in a logbook and repeating this process for eight weeks.
6. Clinical Evaluation:

   - Weekly clinical evaluations will be conducted for mucositis, diarrhea, colitis, flatulence, abdominal distention, and constipation, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) scale (V 4.02) [39]. If necessary, the pediatric oncologist will initiate treatment according to the Oncology service plan.
7. Data Collection:

   * If antibiotics are required or the chemotherapy consolidation phase is completed, participants will be eliminated from the study, and final assessments will be conducted.
   * Data from weekly clinical evaluations, nutritional assessments, and study follow-ups will be recorded in a data collection form (Appendix 8) and entered an electronic Excel database for statistical analysis using STATA 18 by a blinded researcher.

The sample size was calculated based on data from the study by Reyna-Figueroa, which reported a 0% incidence of diarrhea during the administration L. rhamnosus compared to 10% in participants who did not receive probiotics. Using the formula for proportions, with an alpha error of 0.05, 80% power, and estimating a loss rate of 20%, a sample size of 30 participants was determined for each of the four groups.

Statistical analysis A descriptive analysis will be performed using measures of central tendency to understand the characteristics of the studied sample and to determine the type of distribution of each variable using the Kolmogorov-Smirnoff normality test. For quantitative variables, the mean and standard deviation or median with minimum and maximum values will be calculated, depending on the type of distribution and summarized in tabular form; and data graphically represented by boxplot or bars chats as appropriate.

To compare the quantitative variables between the four interventions, a multi-way ANOVA test will be used. For qualitative variables, the chi-squared test will be used to compare the groups, adjusting for the nutritional status of the participants.

The risk of gastrointestinal toxicity and adverse events will be analyzed by the relative risk or Peto's odds ratio and 95% confidence interval. Differences between the interventions will be analyzed using survival analysis with the Kaplan-Meier and Log-Rank tests. Sequencing data will be analyzed using the Qiime2 program, filtered to generate a phylogenetic tree using the Silva database. Corresponding plots will be generated for each taxonomic level. Alpha (intra-group) and Beta (inter-group) diversity will be presented by ordination plots using principal component analysis with the ANCOM program.

Noted that patients who drop out of the study will have their results analyzed up to their last record, and all analyses will be conducted on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 6 years and younger than 17 years with a recent diagnosis of acute lymphoblastic leukemia, confirmed by bone marrow aspirate and interpreted by a pediatric oncologist.
* Participants of both sexes
* Participants receiving treatment at the Oncology Service of the Instituto Nacional de Pediatría.
* Receiving chemotherapy according to national health protocols in the consolidation phase.
* Informed consent
* Informed assent for those older than 8 years.

Exclusion Criteria:

* Allergy to probiotics.
* Consumption of another probiotic
* Enteropathies affecting intestinal absorption (e.g., malabsorption syndrome, short bowel syndrome, intestinal malrotation, chronic nonspecific ulcerative colitis, Crohn's disease).
* Chronic diarrhea (>15 days of duration)
* Presence of mucosal lesions
* Impossibility of enteral feeding
* Renal insufficiency
* Peritoneal dialysis
* Water and electrolyte disorders
* Surgical intestinal bypass (e.g., colostomy, ileostomy)
* Congenital metabolic disorders
* Septicemia
* Body temperature > 38° C
* Received broad-spectrum antibiotics (piperacillin/tazobactam, fourth generation cephalosporins, aminoglycosides, carbapenem and/or metronidazole) within the past 30 days.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevention of Mucositis | 8 weeks
  Inflammation of the oral mucosa and gastrointestinal tract, triggered by the activation of inflammatory cytokines. For the evaluation, the pediatric oncologist will perform the physical examination of the oral cavity and report his findings as follows:
  * Number of participants with mucositis
  * Participants with mucositis will be evaluated with:
  A) The number and location of lesion(s). B) The maximum diameter of the largest lesion in centimeters. C) The severity of lesions
  Grade 1: Mucosal erythema, preserved feeding Grade 2: Focal pseudomembranous ulceration, modified food intake Grade 3: Confluent pseudomembranous ulcers, bleeding with minimal trauma, inability to feed or hydrate.
  Grade 4: Tissue necrosis, significant spontaneous bleeding
Prevention of Diarrhea | 8 weeks
  Increase in stool frequency or a decrease in stool consistency.
  For the evaluation, the pediatric oncologist will question the participant about the characteristics of the bowel movements and perform a physical examination of the abdomen. His findings will be reported as follows: The findings will be recorded as follows:
  * Number of participants with diarrhea
  * Participants with diarrhea will be evaluated with:
  A) Number of bowel movements per day B) Duration of diarrhea in days C) Stool content: None, blood, mocus, fat, food
  D) Classification of the diarrhea episode:
  Grade 1: Fewer than 4 stools per day. Grade 2: 4 to 6 stools per day, requiring intravenous hydration for less than 24 hours.
  Grade 3: More than 7 stools per day, requiring IV hydration for more than 24 hours, and necessitating hospitalization.
  Grade 4: Severe dehydration with hemodynamic consequences, requiring urgent IV hydration.
Prevention of Colitis | 8 weeks
  Inflammation and edema of the intestinal mucosa accompanied by abdominal pain, watery and bloody diarrhea. For the evaluation, the pediatric oncologist and pediatric surgeon, will perform a physical examination, laboratory and imaging studies. Findings will be recorded as follows:
  * Number of participants with colitis
  * Participants with colitis will be assessed with:
  A) Pain intensity using a visual analog scale (0 = no pain to 10 = severe pain).
  B) Location of pain (generalized or in one or more of the 9 abdominal regions) C) Duration of abdominal pain in days
  D) Classification of colitis:
  Grade 1 = asymptomatic Grade 2 = abdominal pain, presence of mucus or blood on evacuation Grade 3 = abdominal pain, fever, changes in evacuation rhythm with ileus or signs of peritoneal irritation.
  Grade 4 = Intestinal perforation, ischemia, hemorrhage, toxic megacolon or intestinal necrosis.
Adverse events (flatulence) | 8 weeks
  Production of intestinal gas mixture that is expelled through the rectum.
  For evaluation, the pediatric oncologist will ask the participant if there has been an increase in the frequency and amount of intestinal gas production during the week, and depending on the characteristics of the abdomen, flatulence will be classified according to the number of gases expelled per day. The findings will be recorded as follows:
  - Number of participants with gas. Absence < 25 gases per day Presence > 25 gases per day
Adverse events (distention) | 8 weeks
  Increased abdominal girth due to excessive gas in the bowel
  For evaluation, the pediatric oncologist will ask the participant if he/she has had an increase in abdominal girth during the week and will measure the abdominal girth using a circumference tape placed around the midpoint between the lower edge of the last rib and the upper edge of the iliac crest without applying pressure and will ask the participant to take a deep breath and at the moment of exhalation the measurement will be taken in centimeters.
Adverse events (constipation) | 8 weeks
  Infrequent bowel movements accompanied by scanty and hard stools. For evaluation, the pediatric oncologist and pediatric surgeon will ask the participant if has had difficulty passing stools during the week and will perform a physical examination. The findings will be recorded as follows:
  * Number of participants with constipation absent = > 1 defecation per day present < 1 defecation per day
  * Participants with constipation will be assessed with:
  A) Frequency of defecation per week B) Length of constipation in days
  C) Classification of constipation:
  Grade 1 = occasional or intermittent symptoms, sporadic use of laxatives, dietary changes, or need for enemas.
  Grade 2 = persistent symptoms with frequent use of laxatives or enemas Grade 3 = symptoms interfere with activities of daily living and require manual bowel movements Grade 4 = risk of death from bowel obstruction or toxic megacolon
Adverse events (vomiting) | 8 weeks
  Violent expulsion of gastric contents by mouth.
  To assess this, the pediatric oncologist will ask the participant if he/she has experienced this during the week. The findings will be recorded as follows:
  * Number of participants who vomited absent present > 1 event per day
  * Participants with vomiting will be assessed with:
  A) Frequency of vomiting per day. B) Duration of vomiting C) Volume of vomiting
  D) Content of vomiting:
  * water
  * blood
  * mucus
  * food

SECONDARY OUTCOMES:
Blood Beta-Lactoglobulin Concentration | 8 weeks
  To determine the functional status of the intestinal wall as a selective barrier to the passage of toxic substances and dietary proteins into the blood (intestinal permeability), the medical oncologist will take a peripheral blood sample by venipuncture and analyze it by sandwich enzyme immunoassay technique for the detection of antibodies against beta-lactoglobulin at the beginning and end of the participant's follow-up. The results will be reported in ng/mL.
Changes in alpha and beta diversity of the intestinal microbiota | 8 weeks
  Gut microbiota, gut microbiome, or gut flora are the microorganisms, including bacteria, archaea, fungi, and viruses, that live in the digestive tracts of animals.The gastrointestinal metagenome is the aggregate of all the genomes of the gut microbiota.The gut is the main location of the human microbiome.The gut microbiota has broad impacts, including effects on colonization, resistance to pathogens, maintaining the intestinal epithelium, metabolizing dietary and pharmaceutical compounds, controlling immune function, and even behavior through the gut-brain axis
Adverse events (fever) | 8 weeks
  Increase in body temperature > 38° C in response to a medical condition.
  For evaluation, the pediatric oncologist will ask about the presence of fever during the week and will take the body temperature with a digital thermometer. The findings will be recorded as follows
  - Number of participants with fever absent < 38 °C present > 38 °C
Adverse events (nausea) | 8 weeks
  Feeling of unpleasantness or intense disgust with proximity to vomiting due to an triggering event.
  To assess this, the pediatric oncologist will ask the participant if he/she is experiencing, or has experienced during the week, a feeling of intense disgust. The findings are recorded as follows
  - Number of participants with nausea absent present

CONTACTS AND LOCATIONS:
Overall Officials: Sara Espinosa-Padilla, Ph.D., Study Director — National Institute of Pediatrics
Locations (1):
- National Institute of Pediatrics, Mexico City, Coyoacan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pui CH, Evans WE. Acute lymphoblastic leukemia. N Engl J Med. 1998 Aug 27;339(9):605-15. doi: 10.1056/NEJM199808273390907. No abstract available. PMID 9718381
- [Background] Pui CH, Campana D, Pei D, Bowman WP, Sandlund JT, Kaste SC, Ribeiro RC, Rubnitz JE, Raimondi SC, Onciu M, Coustan-Smith E, Kun LE, Jeha S, Cheng C, Howard SC, Simmons V, Bayles A, Metzger ML, Boyett JM, Leung W, Handgretinger R, Downing JR, Evans WE, Relling MV. Treating childhood acute lymphoblastic leukemia without cranial irradiation. N Engl J Med. 2009 Jun 25;360(26):2730-41. doi: 10.1056/NEJMoa0900386. PMID 19553647
- [Background] Rivera-Luna R, Velasco-Hidalgo L, Zapata-Tarres M, Cardenas-Cardos R, Aguilar-Ortiz MR. Current outlook of childhood cancer epidemiology in a middle-income country under a public health insurance program. Pediatr Hematol Oncol. 2017 Feb;34(1):43-50. doi: 10.1080/08880018.2016.1276236. Epub 2017 Mar 13. PMID 28287336
- [Background] Moricke A, Zimmermann M, Valsecchi MG, Stanulla M, Biondi A, Mann G, Locatelli F, Cazzaniga G, Niggli F, Arico M, Bartram CR, Attarbaschi A, Silvestri D, Beier R, Basso G, Ratei R, Kulozik AE, Lo Nigro L, Kremens B, Greiner J, Parasole R, Harbott J, Caruso R, von Stackelberg A, Barisone E, Rossig C, Conter V, Schrappe M. Dexamethasone vs prednisone in induction treatment of pediatric ALL: results of the randomized trial AIEOP-BFM ALL 2000. Blood. 2016 Apr 28;127(17):2101-12. doi: 10.1182/blood-2015-09-670729. Epub 2016 Feb 17. PMID 26888258
- [Background] Barry E, Alvarez JA, Scully RE, Miller TL, Lipshultz SE. Anthracycline-induced cardiotoxicity: course, pathophysiology, prevention and management. Expert Opin Pharmacother. 2007 Jun;8(8):1039-58. doi: 10.1517/14656566.8.8.1039. PMID 17516870
- [Background] Schmiegelow K, Muller K, Mogensen SS, Mogensen PR, Wolthers BO, Stoltze UK, Tuckuviene R, Frandsen T. Non-infectious chemotherapy-associated acute toxicities during childhood acute lymphoblastic leukemia therapy. F1000Res. 2017 Apr 7;6:444. doi: 10.12688/f1000research.10768.1. eCollection 2017. PMID 28413626
- [Background] Gorschluter M, Marklein G, Hofling K, Clarenbach R, Baumgartner S, Hahn C, Ziske C, Mey U, Heller R, Eis-Hubinger AM, Sauerbruch T, Schmidt-Wolf IG, Glasmacher A. Abdominal infections in patients with acute leukaemia: a prospective study applying ultrasonography and microbiology. Br J Haematol. 2002 May;117(2):351-8. doi: 10.1046/j.1365-2141.2002.03434.x. PMID 11972517
- [Background] Inaba H, Pei D, Wolf J, Howard SC, Hayden RT, Go M, Varechtchouk O, Hahn T, Buaboonnam J, Metzger ML, Rubnitz JE, Ribeiro RC, Sandlund JT, Jeha S, Cheng C, Evans WE, Relling MV, Pui CH. Infection-related complications during treatment for childhood acute lymphoblastic leukemia. Ann Oncol. 2017 Feb 1;28(2):386-392. doi: 10.1093/annonc/mdw557. PMID 28426102
- [Background] Ribeiro ILA, Limeira RRT, Dias de Castro R, Ferreti Bonan PR, Valenca AMG. Oral Mucositis in Pediatric Patients in Treatment for Acute Lymphoblastic Leukemia. Int J Environ Res Public Health. 2017 Nov 28;14(12):1468. doi: 10.3390/ijerph14121468. PMID 29182564
- [Background] Raja RA, Schmiegelow K, Albertsen BK, Prunsild K, Zeller B, Vaitkeviciene G, Abrahamsson J, Heyman M, Taskinen M, Harila-Saari A, Kanerva J, Frandsen TL; Nordic Society of Paediatric Haematology and Oncology (NOPHO) group. Asparaginase-associated pancreatitis in children with acute lymphoblastic leukaemia in the NOPHO ALL2008 protocol. Br J Haematol. 2014 Apr;165(1):126-33. doi: 10.1111/bjh.12733. Epub 2014 Jan 15. PMID 24428625
- [Background] Hudson MM, Ness KK, Gurney JG, Mulrooney DA, Chemaitilly W, Krull KR, Green DM, Armstrong GT, Nottage KA, Jones KE, Sklar CA, Srivastava DK, Robison LL. Clinical ascertainment of health outcomes among adults treated for childhood cancer. JAMA. 2013 Jun 12;309(22):2371-2381. doi: 10.1001/jama.2013.6296. PMID 23757085
- [Background] Strauss AJ, Su JT, Dalton VM, Gelber RD, Sallan SE, Silverman LB. Bony morbidity in children treated for acute lymphoblastic leukemia. J Clin Oncol. 2001 Jun 15;19(12):3066-72. doi: 10.1200/JCO.2001.19.12.3066. PMID 11408503
- [Background] Zawitkowska J, Lejman M, Zaucha-Prazmo A, Drabko K, Plonowski M, Bulsa J, Romiszewski M, Mizia-Malarz A, Koltan A, Derwich K, Karolczyk G, Ociepa T, Cwiklinska M, Trelinska J, Owoc-Lempach J, Niedzwiecki M, Kiermasz A, Kowalczyk J. Grade 3 and 4 Toxicity Profiles During Therapy of Childhood Acute Lymphoblastic Leukemia. In Vivo. 2019 Jul-Aug;33(4):1333-1339. doi: 10.21873/invivo.11608. PMID 31280227
- [Background] Boussios S, Pentheroudakis G, Katsanos K, Pavlidis N. Systemic treatment-induced gastrointestinal toxicity: incidence, clinical presentation and management. Ann Gastroenterol. 2012;25(2):106-118. PMID 24713845
- [Background] Ruiz-Esquide G, Nervi B, Vargas A, Maiz A. [Treatment and prevention of cancer treatment related oral mucositis]. Rev Med Chil. 2011 Mar;139(3):373-81. Epub 2011 Aug 25. Spanish. PMID 21879172
- [Background] Moscardo Guilleme C, Fernandez Delgado R, Sevilla Navarro J, Astigarraga Aguirre I, Rives Sola S, Sanchez de Toledo Codina J, Fuster Soler JL, Parra Ramirez L, Molina Garicano J, Gonzalez Martinez B, Madero Lopez L. [Update on L-asparaginase treatment in paediatrics]. An Pediatr (Barc). 2013 Nov;79(5):329.e1-329.e11. doi: 10.1016/j.anpedi.2013.03.015. Epub 2013 May 31. Spanish. PMID 23727426
- [Background] El-Mahallawy HA, El-Din NH, Salah F, El-Arousy M, El-Naga SA. Epidemiologic profile of symptomatic gastroenteritis in pediatric oncology patients receiving chemotherapy. Pediatr Blood Cancer. 2004 Apr;42(4):338-42. doi: 10.1002/pbc.10394. PMID 14966830
- [Background] Maroun JA, Anthony LB, Blais N, Burkes R, Dowden SD, Dranitsaris G, Samson B, Shah A, Thirlwell MP, Vincent MD, Wong R. Prevention and management of chemotherapy-induced diarrhea in patients with colorectal cancer: a consensus statement by the Canadian Working Group on Chemotherapy-Induced Diarrhea. Curr Oncol. 2007 Feb;14(1):13-20. doi: 10.3747/co.2007.96. PMID 17576459
- [Background] Ahern PP, Maloy KJ. Understanding immune-microbiota interactions in the intestine. Immunology. 2020 Jan;159(1):4-14. doi: 10.1111/imm.13150. Epub 2019 Nov 27. PMID 31777071
- [Background] Icaza-Chavez ME. [Gut microbiota in health and disease]. Rev Gastroenterol Mex. 2013 Oct-Dec;78(4):240-8. doi: 10.1016/j.rgmx.2013.04.004. Epub 2013 Nov 28. Spanish. PMID 24290319
- [Background] Hawrelak JA, Myers SP. The causes of intestinal dysbiosis: a review. Altern Med Rev. 2004 Jun;9(2):180-97. PMID 15253677
- [Background] Forsgard RA, Marrachelli VG, Korpela K, Frias R, Collado MC, Korpela R, Monleon D, Spillmann T, Osterlund P. Chemotherapy-induced gastrointestinal toxicity is associated with changes in serum and urine metabolome and fecal microbiota in male Sprague-Dawley rats. Cancer Chemother Pharmacol. 2017 Aug;80(2):317-332. doi: 10.1007/s00280-017-3364-z. Epub 2017 Jun 23. PMID 28646338
- [Background] Hakim H, Dallas R, Wolf J, Tang L, Schultz-Cherry S, Darling V, Johnson C, Karlsson EA, Chang TC, Jeha S, Pui CH, Sun Y, Pounds S, Hayden RT, Tuomanen E, Rosch JW. Gut Microbiome Composition Predicts Infection Risk During Chemotherapy in Children With Acute Lymphoblastic Leukemia. Clin Infect Dis. 2018 Aug 1;67(4):541-548. doi: 10.1093/cid/ciy153. PMID 29518185
- [Background] Touchefeu Y, Montassier E, Nieman K, Gastinne T, Potel G, Bruley des Varannes S, Le Vacon F, de La Cochetiere MF. Systematic review: the role of the gut microbiota in chemotherapy- or radiation-induced gastrointestinal mucositis - current evidence and potential clinical applications. Aliment Pharmacol Ther. 2014 Sep;40(5):409-21. doi: 10.1111/apt.12878. Epub 2014 Jul 11. PMID 25040088
- [Background] Reyna-Figueroa J, Barron-Calvillo E, Garcia-Parra C, Galindo-Delgado P, Contreras-Ochoa C, Lagunas-Martinez A, Campos-Romero FH, Silva-Estrada JA, Limon-Rojas AE. Probiotic Supplementation Decreases Chemotherapy-induced Gastrointestinal Side Effects in Patients With Acute Leukemia. J Pediatr Hematol Oncol. 2019 Aug;41(6):468-472. doi: 10.1097/MPH.0000000000001497. PMID 31033786
- [Background] Wei D, Heus P, van de Wetering FT, van Tienhoven G, Verleye L, Scholten RJ. Probiotics for the prevention or treatment of chemotherapy- or radiotherapy-related diarrhoea in people with cancer. Cochrane Database Syst Rev. 2018 Aug 31;8(8):CD008831. doi: 10.1002/14651858.CD008831.pub3. PMID 30168576
- [Background] Alexander JL, Wilson ID, Teare J, Marchesi JR, Nicholson JK, Kinross JM. Gut microbiota modulation of chemotherapy efficacy and toxicity. Nat Rev Gastroenterol Hepatol. 2017 Jun;14(6):356-365. doi: 10.1038/nrgastro.2017.20. Epub 2017 Mar 8. PMID 28270698
- [Background] Redman MG, Ward EJ, Phillips RS. The efficacy and safety of probiotics in people with cancer: a systematic review. Ann Oncol. 2014 Oct;25(10):1919-1929. doi: 10.1093/annonc/mdu106. Epub 2014 Mar 11. PMID 24618152
- [Background] Lu D, Yan J, Liu F, Ding P, Chen B, Lu Y, Sun Z. Probiotics in preventing and treating chemotherapy-induced diarrhea: a meta-analysis. Asia Pac J Clin Nutr. 2019;28(4):701-710. doi: 10.6133/apjcn.201912_28(4).0005. PMID 31826366
- [Background] Rodriguez JM, Murphy K, Stanton C, Ross RP, Kober OI, Juge N, Avershina E, Rudi K, Narbad A, Jenmalm MC, Marchesi JR, Collado MC. The composition of the gut microbiota throughout life, with an emphasis on early life. Microb Ecol Health Dis. 2015 Feb 2;26:26050. doi: 10.3402/mehd.v26.26050. eCollection 2015. PMID 25651996
- [Background] Van den Nieuwboer M, Brummer RJ, Guarner F, Morelli L, Cabana M, Claasen E. The administration of probiotics and synbiotics in immune compromised adults: is it safe? Benef Microbes. 2015 Mar;6(1):3-17. doi: 10.3920/BM2014.0079. PMID 25304690
- See also: Cancer Stat Facts: Leukemia — https://seer.cancer.gov/statfacts/html/leuks.html